CLINICAL TRIAL: NCT07199075
Title: Fusion Rate of Anterior Lumbar Interbody Fusion and Extreme Lateral Interbody Fusion Using Titanium Cages Filled With Stand-alone Fibergraft in Lumbar Spinal Fusion
Brief Title: Rate of Bone Union After Surgery With Stand-alone Fibergraft
Acronym: Fibergraft
Status: Not yet recruiting | Type: Observational
Sponsor: AO Innovation Translation Center (Other)
Responsible Party: Sponsor
Other Study IDs: Fibergraft
Record Dates: First submitted 2025-09-22; First posted 2025-09-30 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: Spine Degeneration; Spine Disorder; Spine Pain; Spine Fusion; Spine Fusion for Degenerative Spine Disease; Nerve Root Compress;Lumbosac; Spondylolisthesis
MeSH Terms: conditions — Spinal Diseases; Spondylolisthesis | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Questionnaires — Questionnaires
  * Oswestry Disability Index (ODI)
  * Pain NRS lower back and (wors side) leg
  * EQ-5D-3L
Radiation: Computer Tomography — One additional CT scan is performed for some patients

SUMMARY:
Some people have back problems caused by degenerative conditions or instability of the spine (eg. Spondylolisthesis). These problems can lead to pain, nerve issues, or difficulties in walking. A common treatment is a type of back surgery called lumbar interbody fusion, which helps stabilize the spine.

At the St. Maartenskliniek in the Netherlands, doctors have been using a special material called Fibergraft Bioactive Glass Putty for such surgeries since 2023. This material helps bones grow and heal, and it's placed inside the spine without needing extra bone from another part of the body.

This study will look at how well this material works by evaluating how many patients' bones successfully healed after surgery using this material. It will also look at how patients feel and recover after the procedure

DETAILED DESCRIPTION:
Lumbar interbody fusion is an established procedure for patients with lumbar degenerative conditions and spondylolisthesis, with symptoms of pain, radiculopathy, and/or myelopathy. Completion of fusion, ie, union, of an intended motion segment remains a desirable endpoint of spinal fusion, supported by the observations that pseudoarthrosis, ie, nonunion, following spinal fusion is correlated with poorer patient outcomes.

Iliac crest bone autograft is considered the gold standard for spinal fusion with excellent fusion rates and clinical outcomes. However, its clinical use has been restricted due to limited availability of harvestable bone, donor-site morbidity, increased surgical time, and the need for additional surgical staff and associated costs. As a result, there has been great interest in the search for bone graft substitutes to replace or reduce the amount of autograft, which will lower the risks associated with the harvesting procedure while still providing a favorable environment for a solid fusion. A wide range of synthetic bone grafts have been explored, including ceramics, bioactive glasses, and polymer-based compounds.

Although bioactive glasses have been used in spinal fusion for three decades, literature on them is dispersed over the wide array of bioactive glasses investigated and numerous small clinical studies. There is marked variability in these studies in terms of the patient population, indications, procedures performed, single- vs multi-level procedures, types of bioactive glasses, use of autografts, duration of follow-up (FU), and methods to determine fusion status. It is therefore difficult to draw conclusions on the optimal bioactive glass for a particular application. Nonetheless, the current literature suggests that bioactive glasses may be effective as bone graft extenders when combined with autograft to promote spinal fusion, yielding at least noninferior fusion rates when compared with autograft alone. There is limited data regarding the effectiveness of bone glasses as standalone bone graft substitutes or in interbody fusion procedures.

This single-center study to be conducted at the St. Maartenskliniek, the Netherlands, aims to address this knowledge gap. Since 2023, the hospital has consistently used Fibergraft Bioactive Glass (BG) Putty, a product from the FIBERGRAFTTM Bioactive Bone Graft Substitute family (Johnson & Johnson MedTech), as standalone cage fillers for anterior lumbar interbody fusion (ALIF) and extreme lateral interbody fusion (XLIF). This provides an opportunity for a case series to determine the fusion rate for bioactive glass as a standalone bone graft substitute in lumbar interbody fusion.

ELIGIBILITY:
Inclusion Criteria:

* Adults ≥ 18 years old
* Diagnosed with the following lumbar spine disorders: foraminal nerve root compression, isthmic spondylolisthesis, and short-segment (1-2 levels) deformity.
* Undergone primary surgery of ALIF or XLIF using titanium cages filled with standalone Fibergraft and with the following criteria fulfilled (ie, the index surgery):

  * ALIF (up to 2 levels) as either standalone (ie, no posterior procedure) or as an anterior first procedure with posterior procedure as a second procedure.
  * XLIF (up to 2 levels) as an anterior first procedure with posterior procedure as a second procedure.
* Consenting to have CT scans taken to allow assessment of fusion status at 12-24 months post index surgery

  * This criterion is applicable to patients who have not undergone revision surgery.
  * For patients who have undergone revision surgery due to any reason other than nonunion, which typically occurs within 1 year of the index surgery, this criterion is only applicable if it is possible to obtain the CT scan within 12-24 months of the index surgery. If no CT scan can be taken during this window, the patient does not need to undergo the CT scan; in such cases, the CT scan that has been taken as part of the standard of care before the revision surgery will be retrospectively retrieved to assess the fusion status at the time of the revision surgery.
  * This criterion is not applicable to patients who underwent revision surgery due to nonunion, which typically occurs 1 year after the index surgery; these patients do not need to undergo the CT scan. In such cases, the CT scan that has been taken as part of the standard of care before the revision surgery will also be retrospectively retrieved to assess and grade the fusion status at the time of the revision surgery.
* Ability to provide informed consent according to the IRB/EC defined and approved procedures

Exclusion Criteria:

* Revision surgery
* Standalone XLIF
* Posterior lumbar interbody fusion
* Diagnosis of fractures, malignancies, ankylosing spondylitis, or acute cauda equina syndrome
* Diagnosis of Parkinson's disease
* Body mass index > 35kg/m2

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with spinal degenerative deseases from the St Mateenskliniek
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2025-10-31 (Estimated); Primary Completion 2026-05-30 (Estimated); Study Completion 2026-05-30 (Estimated)

PRIMARY OUTCOMES:
Interbody fusion status | 12months to 24th months after index surgery
  The primary outcome measure is the interbody fusion status determined by a regular lumbar spine CT scan protocol without additional radiation or contrast agents. The patients will be evaluated with one CT-scan within a window of 12 to 24 months postsurgery. The Bridwell Interbody Fusion Grading Classification will be used to assess fusion status for each intended segment.

SECONDARY OUTCOMES:
Oswestry Disability Index (ODI) | Before the index surgery and 12-24months post index surgery
  The level of disability will be measured using the ODI . The ODI is a self-administered questionnaire divided into ten sections designed to assess limitations of various activities of daily living. Each section is scored on a 0-5 scale, with 5 representing the greatest disability. The index is calculated by dividing the sum of the scores by the total possible score, which is then multiplied by 100 and expressed as a percentage. The preoperative ODI will be retrospectively collected via medical records, and patients will fill out the ODI at the 12-24 months visit.
General back pain and (worse side) leg pain | Before the index surgery and 12-24 months after the index surgery
  General back pain and (worse side) leg pain will be measured by the patients on an NRS of 0 to 10, with 0 representing no pain and 10 the worst imaginable pain.
  Preoperative pain NRS will be retrospectively collected via medical records, and patients will fill out pain NRS at the 12-24 months visit.
The EuroQoL-5 Dimension | Before the index surgery and 12-24months after the index surgery
  The EQ-5D is a generic measure of self-reported health developed by the EuroQol Group. It measures five dimensions for describing health states: mobility, usual activities, self-care, pain and discomfort, and anxiety and depression. The questionnaire is comprised of two parts. The first part is the EQ-5D descriptive system, in which individuals are asked to indicate the level of problem they experience on each of the five dimensions. The second part is the EQ Visual Analogue Scale, which captures the individual's overall health on a scale from 0 (worst health imaginable) to 100 (best health imaginable). For this study, the EQ-5D-3L (3 levels) version will be used.
  Preoperative EQ-5D-3L will be retrospectively collected via medical records, and patients will fill out EQ-5D-3L at the 12-24 months visit.
Patient's overall satisfaction | 12months to 24th months after the index surgery
  Patients' overall satisfaction with the treatment will be measured on a 7-point Likert scale at the 12-24 months visit.
  * Extremely satisfied
  * Very satisfied
  * Somewhat satisfied
  * Mixed (approximately equal satisfaction and dissatisfaction)
  * Somewhat dissatisfied
  * Very dissatisfied
  * Extremely dissatisfied
Complications | From after the index surgery until the visit at 12months to 24months after the index surgery
  The following AEs/complications are of particular interest to the study. The dates when they occur and their treatments (reoperation, medical treatment, or no interventions) will be documented:
  * Dural tear (if the patient has undergone posterior procedure)
  * Persistent radiculopathy
  * Sensory deficit
  * Motor deficit
  * Persistent back pain
  * Cauda syndrome (if the patient has undergone posterior procedure)
  * Retrograde ejaculation (for male patients)
  * Vascular injury (if the patient has undergone anterior procedure)
  * Hardware failure
  * Pseudoarthrosis
  * Persistent wound leakage
  * Surgical wound infection (superficial)
  * Surgical wound infection (deep)
  * Deep vein thrombosis
  * Pulmonary embolism
  * Pneumonia
  * Urinary tract infection
  * Other, specify
  In addition to postoperative complications, several radiographic findings and the date of detection on images will also be recorded:
  • Cage subsidence
  * If yes, levels of cage subsidence (multiple answers possible): T12-L1 to L5-S1
  * For
Reoperations | From after the index surgery until the 12months to 24months visit after the index surgery
  Any reoperation of the index levels and the adjacent levels, such as revision, removal of implants, and supplemental fixation, will be documented

CONTACTS AND LOCATIONS:
Locations (1):
- St Mateenskliniek, Ubbergen, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
All IPD collected for this study